CLINICAL TRIAL: NCT04358341
Title: Phase II Study of Pegliposomal Doxorubicin and 5-fluorouracil Compared With Irinotecan as Second Line Therapy for Metastatic Gastric Cancer.
Brief Title: Pegliposomal Doxorubicin and 5-fluorouracil as Second Line Therapy for Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Asso. Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO205
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Gastric Cancer
Keywords: Pegliposomal Doxorubicin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Doxorubicin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan alone (Active Comparator): 150 mg/m2 iv drip d1; Repeat every 14 days.
  Interventions: Drug: Irinotecan
- Pegliposomal Doxorubicin and 5-FU (Experimental): Pegliposomal Doxorubicin: 25mg/m2 iv drip d1; 5FU 400mg/m2 iv bolus and 2400 mg/m2 civ 46h d1; Repeat every 14 days.
  Interventions: Drug: DOXOrubicin Liposome Injection; Drug: 5fluorouracil

INTERVENTIONS:
Drug: Irinotecan — 150 mg/m2 ivdrip every 14 days
  Other Names: CPT-11
  Arms: Irinotecan alone
Drug: DOXOrubicin Liposome Injection — 25 mg/m2 ivdrip every 14 days
  Other Names: Pegliposomal Doxorubicin
  Arms: Pegliposomal Doxorubicin and 5-FU
Drug: 5fluorouracil — 400mg/m2 iv bolus and 2400 mg/m2 civ 46h every 14 days
  Other Names: 5-FU
  Arms: Pegliposomal Doxorubicin and 5-FU

SUMMARY:
For second-line chemotherapy for metastatic gastric cancer, single-agent irinotecan is the standard treatment. Anthracyclines are active but lack well designed investigations. The combination of epirubicin, fluorouracil and cisplatin (or oxaliplatin) are widely used in Europe. However, traditional anthracyclines are more cardiotoxic; and (Pegliposomal Doxorubicin) PLD, as a new liposome dosage form of doxorubicin, has better cardiac safety. Therefore, we designed this phase II trial with PLD and 5-Fu to compare irinotecan monotherapy in the second-line treatment.

DETAILED DESCRIPTION:
Patients with metastatic gastric cancer failed to first-line therapy will be radomized to arm A with PLD and 5-Fu and arm B with irinotecan single agent therapy. Both regimens will be treated every 2 weeks until disease progression or untolerable toxicity. Efficacy will be assessed every 3 cycles and safety will be evaluated every cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old;
2. Metastatic gastric cancer progressed on first-line treatment;
3. Expected survival time ≥ 3 months;
4. At least one evaluable target lesion according to the solid tumor evaluation criteria (RECIST) version 1.1;
5. ECOG PS 0~2;
6. Adequate bone marrow function reserve: white blood cell count ≥ 3.0 × 10*9 / L, neutrophil count ≥ 1.5 × 10*9/ L; platelet count ≥ 100 ×10*9/ L; hemoglobin ≥ 90 g / L;
7. Adequate liver and renal function reserve: AST and ALT ≤ 2.5 times the upper limit of normal value, total bilirubin ≤ 2 times the upper limit of normal value; serum creatinine ≤ 1.5 times the upper limit of normal value;
8. LVEF ≥ 55 %;
9. Be able to understand the research process, volunteer to participate in the study, and sign an informed consent form.

Exclusion Criteria:

1. Patients known to be allergic to active or other components of chemotherapeutic drugs;
2. Patients who have been treated with PLD or irinotecan in the past;
3. According to the researcher's judgment, other anti-tumor treatments such as radiotherapy and surgical resection are required during chemotherapy;
4. Those who are not expected to be able to tolerate chemotherapy with severe heart disease or discomfort;
5. d-MMR or MSI-H or Her-2 overexpression;
6. Severe or uncontrolled infections or diabetes;
7. History of other malignacis in the past 5 years (except for cured cervical carcinoma in situ or basal cell carcinoma of the skin);
8. Participated in other clinical trials within 4 weeks prior to the start of the study;
9. Pregnant or lactating women, or women of childbearing age who refuse to take effective contraception during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 24 weeks
  Percentage of subjects with tumor shrinkage reaching complete response (CR), partial response (PR) and disease stabilization (SD).

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 weeks
  Percentage of subjects with tumor shrinkage reaching complete response (CR) and partial remission (PR).
Progression-Free Survival (PFS) | 1 year
  PFS is defined as the time from the date of randomization to the date of the first documentation of progressive disease or date of death, whichever occurs first. For target lesions (TL), PD was defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD) of TLs, taking as a reference the smallest SLD recorded since the treatment started, or the appearance of one or more lesions. For non-target lesions (NTL), PD was defined as an unequivocal progression of existing NTLs. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up.
Overall Survival (OS) | 2 years
  OS is defined as the time from the date of randomization to the date of death due to any cause. Participants were censored at the last date of tumor measurement, the last date in the study drug log or the date of last follow-up.
Treatment associated toxicities | 2 years
  According to WHO CTC 3.0
EORTC Quality of Life Questionnaire-Stomach Cancer Specific (QLQ STO22) Questionnaire Scores | 2 years
  The QLQ-STO22 is a gastric cancer quality of life questionnaire. There are 22 questions concerning disease, treatment related symptoms, side effects, dysphagia, nutritional aspects, and questions about the emotional problems of gastric cancer (dysphagia, pain, reflux, eating restrictions, anxiety, dry mouth, body image, and hair loss). The questions are grouped into five scales and 4 single items which are related to the symptoms of the disease. Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Jian Xiao, Guangzhou, Guangdong, China